CLINICAL TRIAL: NCT04038619
Title: Fecal Microbiota Transplantation (FMT) for Immune-Checkpoint Inhibitor Induced-Diarrhea/Colitis in Genitourinary Cancer Patients
Brief Title: Fecal Microbiota Transplantation in Treating Immune-Checkpoint Inhibitor Induced-Diarrhea or Colitis in Genitourinary Cancer Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0663; NCI-2019-02660 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0663 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-07-26; First posted 2019-07-31 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Colitis; Diarrhea; Malignant Genitourinary System Neoplasm; Melanoma; Lung Cancer; Ovarian Cancer; Uterine Cancer; Breast Cancer; Cervical Cancer
MeSH Terms: conditions — Colitis; Diarrhea; Urogenital Neoplasms; Melanoma; Lung Neoplasms; Ovarian Neoplasms; Uterine Neoplasms; Breast Neoplasms; Uterine Cervical Neoplasms | interventions — Fecal Microbiota Transplantation; Loperamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (loperamide, colonoscopy, FMT) (Experimental): Patients receive loperamide PO. After 4 hours, patients undergo FMT via colonoscopy over 15-30 minutes.
  Interventions: Procedure: Fecal Microbiota Transplantation; Drug: Loperamide

INTERVENTIONS:
Procedure: Fecal Microbiota Transplantation — Undergo FMT via colonoscopy
  Other Names: Fecal Material Transplantation; Fecal Transplantation; FMT; Poo Transplant; Poop Transplant; Stool Transplant
Drug: Loperamide — Given PO

SUMMARY:
This trial studies how well fecal microbiota transplantation works in treating diarrhea or colitis (inflammation of the intestines) that is caused by certain types of medications (called immune-checkpoint inhibitors) in patients with genitourinary cancer. Fecal microbiota transplantation may effectively reduce the incidence of immune checkpoint inhibitor-induced diarrhea/colitis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

* To assess the safety and tolerability of fecal microbiota transplantation (FMT).
* To assess the efficacy of FMT for clinical remission/response of immune-related diarrhea/colitis.

SECONDARY OBJECTIVES:

- To measure the recurrence rate after achieving clinical remission/response of immune-related diarrhea/colitis.

EXPLORATORY OBJECTIVES:

* To assess the efficacy of FMT to achieve endoscopic remission of immune-related diarrhea/colitis.
* To assess the efficacy of FMT to achieve histological remission of immune-related diarrhea/colitis.
* To assess the efficacy of FMT on recurrence of immune-related diarrhea/colitis after resumption of immune checkpoint inhibitors (ICPI).
* To assess immunological, molecular and microbiome changes in tissue/blood/stool.

To study the efficacy and/ or benefit of PuraStat gel in the healing of mucosal ulcers and its hemostatic effect on bleeding lesions

OUTLINE:

Patients receive loperamide orally (PO). After 4 hours, patients undergo FMT via colonoscopy over 15-30 minutes.

After completion of study treatment, patients are followed up at 2, 4, and 8 weeks, and then at 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of any type of genitourinary (kidney, bladder and prostate), melanoma, non-melanoma skin cancer, lung, head & neck, sarcoma/lymphoma, gastrointestinal system (luminal GI, hepatobiliary, pancreas), gynecology system (ovarian, uterine, cervical), and breast malignancies
2. Treatment with any ICPI agent(s)
3. Participants with new onset of ≥ grade 2 ICPI-induced diarrhea and/or colitis symptoms based on the Common Terminology Criteria for Adverse Events (CTCAE) version 5 within 45 days prior to date of FMT treatment without involvement of non- GI toxicity
4. Participants with a history of steroid use before FMT can be allowed if last dose was > 30 days prior to FMT treatment or treatment duration was for <7 days beyond one week prior to FMT treatment
5. Participants with a history of immunosuppressant (Infliximab, Vedolizumab etc) use before FMT can be allowed if last dose was administered ≥ 3 months prior to FMT treatment when used for the treatment of conditions other than for ICI- induced GI toxicities (e.g., Infliximab is used in the treatment of Crohn's disease, rheumatoid arthritis, plaque psoriasis, and Vedolizumab is used in treating ulcerative colitis)
6. No concern for active concomitant GI infection at the time of initiation of protocol therapy as confirmed by stool tests or as per the treating physician based on clinical presentation
7. Patient has been cleared for enrollment by Infectious Diseases consultant or treating physician if positive infection workup or screening tests (e.g., lifelong positive T-spot due to BCG inoculation, chronic colonization) prior to initiation of protocol therapy and/ or imaging (e.g. CXR, CT CAP etc) confirms the absence of active infections (e.g. TB) within 60 days prior to initiation of protocol therapy
8. Ability to understand and willingness to sign an informed consent form
9. Life expectancy > 6 months

Exclusion Criteria

1. Age younger than 18 years
2. Participants with persistent GI infection confirmed with positive stool test(s) despite completing 5 days of antibiotics prior to initiation of protocol therapy
3. History of inflammatory bowel disease, and/or radiation enteritis or colitis with active disease status at the time of study treatment initiation
4. Pregnant and breastfeeding women
5. Women who have positive urine or serum pregnancy test or refuse to do pregnancy test unless last menstrual cycle was > 1 year prior to consent and/ or clear documentation states that participant is peri- or post-menopausal or there has been recent supporting objective evidence of 'no pregnancy' status (e.g. blood or imaging) within 30 days prior to date of study treatment
6. Immunosuppressive treatment at onset of ICPI-induced diarrhea/colitis
7. Any medical conditions (e.g. severe heart failure, brain hemorrhage, septic shock, etc.) that are high risk for colonoscopy procedure by the assessment of the study PI or Co-PIs.
8. Participants who develop concurrent non-GI toxicity at the time of study treatment
9. Donors at risk for monkeypox infection and/ or exposure as determined by a questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of fecal microbiota transplantation (FMT)-related adverse events | Up to 3 months post-FMT
  Assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5. All events are recorded with grade and attribution to FMT.
Clinical response/remission of immune-related diarrhea/colitis | At 2 weeks post-FMT
  Clinical remission of immune related events defined as improvement of symptoms of grade 1 or lower within 2 weeks post-FMT. Clinical partial response of immune related diarrhea/colitis defined as improvement of diarrhea/colitis to a lower grade than the initial presentation but not meeting criteria of clinical remission at 2 week post-FMT time point.

SECONDARY OUTCOMES:
Recurrent immune-related diarrhea/colitis within 3 months post-FMT after initially achieving clinical remission/response | Up to 3 months post-FMT
  Recurrent immune-related diarrhea colitis events occurring post-FMT are recorded throughout the follow-up period.

OTHER OUTCOMES:
Endoscopic remission (Mayo Clinic sub-score 0-1) of immune-related diarrhea/colitis | At 4 weeks and 8 weeks post-FMT
  Endoscopic remission is defined as Mayo Clinic endoscopic subscore 0 or 1 (absence of ulcers, with or without mild erythema, friability and decreased vascular pattern).
Histological remission (resolution of active inflammation) of immune-related diarrhea/colitis | At 8 weeks post-FMT
  Histological remission is defined resolution of active inflammation on biopsy sample.
Recurrent immune-related diarrhea/colitis following FMT and immune checkpoint inhibitors (ICPI) resumption within 6 months of ICPI resumption | Up to 6 months after restarting ICPI
  Recurrent immune-related diarrhea colitis events occurring post-FMT will be recorded throughout the follow-up period.
Measure immunological measures (including levels of cytokines (IL-6, 17, TNF, etc.) in tissue/blood/stool samples | Up to 3 months
  Blood, stool, and colon tissues will be collected from at each scheduled time point. Markers of interest for immunological and biological profiles include levels of cytokines (IL-6, 17, TNF, etc). Special attention will focus on Bacteroidetes, Akkermansia, and Blautia.
Frequencies of immune cells (CD4/8 T cells, regulatory T cells [Treg], macrophages, etc.) in tissue/blood/stool samples | Up to 3 months
  Blood, stool, and colon tissues will be collected from at each scheduled time point. Markers of interest for immunological and biological profiles include frequencies of immune cells (CD4/8 T cells, Treg, macrophages, etc). Special attention will focus on Bacteroidetes, Akkermansia, and Blautia.

CONTACTS AND LOCATIONS:
Overall Officials: Yinghong Wang, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org